CLINICAL TRIAL: NCT03088332
Title: Prospective Multicenter Study to Evaluate the Efficacy and Results of Endoscopic Gastroplasty Performed Using Overstitch in Patients With Class I and II Obesity.
Brief Title: Evaluating the Efficacy and Results of Endoscopic Gastroplasty Performed Using Overstitch in Patients With Obesity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Clinic and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1854540
Record Dates: First submitted 2017-03-06; First posted 2017-03-23 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic gastroplasty (Experimental): Make a gastric tube similar to that obtained in surgical gastroplication however it will be created using intragastric endoscopic sutures.
  Interventions: Procedure: Endoscopic gastroplasty

INTERVENTIONS:
Procedure: Endoscopic gastroplasty — Vertical endoscopic gastroplasty

SUMMARY:
Obesity is a chronic disease that has grown to epidemic characteristics in Brazil and around the world in recent years. Treatment for patients with class III or class II obesity with comorbidities is already well established, with bariatric surgery being the best option. However, there is no consensus as to the best treatment for cases of class I and class II obesity without comorbidities. The objective of this research will be to make a gastric tube similar to that obtained in surgical gastroplication however it will be created using intragastric endoscopic sutures. The procedures will be performed at the Endoscopy Service of the Mario Covas Hospital in São Paulo, SP. Data collection will be performed at the same location.

DETAILED DESCRIPTION:
The objective of this research will be to make a gastric tube similar to that obtained in surgical gastroplication however it will be created using intragastric endoscopic sutures. The secondary objective will be to correlate demographic, endoscopic and laboratory data with the results of this procedure.

Patients and Methods: Patients with class I obesity with or without comorbidities and patients with class II obesity without comorbidities, irrespective of gender and ethnic background, from the state of São Paulo and other states of the country will be submitted to vertical endoscopic gastroplasty. The procedures will be performed at the Endoscopy Service of the Mario Covas Hospital in São Paulo, SP. Data collection will be performed at the same location.

Information will be obtained during the outpatient follow-up at the Hospital Mario Covas including demographic (gender, age), clinical (height, weight, time after procedure, systemic arterial hypertension, diabetes, dyslipidemia, smoking, alcohol consumption) and operative data (complications).

Preparation for the procedure: All the exams will be performed at the Hospital Mario Covas after the patients have fasted for at least 8 hours. The procedure will begin with the patient in left lateral decubitus under general anesthesia performed by an anesthesiologist. Endoscopic sutures will be performed using 2-0 prolene thread until a tubular-shaped stomach is formed similar to a vertical gastrectomy.

Recovery after the procedure: After the procedure and recovery from anesthesia, all patients will be discharged but only together with a companion. All patients will receive guidance and will remain in touch with a physician to report any adverse signs or symptoms.

Outcomes Primary outcome: To confirm the efficacy of endoscopic sutures in the primary treatment of obesity.

Secondary outcome: To evaluate the use of the endoscopic sutures in relation to demographic data.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 and < 36 with or without comorbidities
* BMI > 36 and < 40 without comorbidities

Exclusion Criteria:

* Prior gastric surgery
* Use of anticoagulants
* Psychiatric disorders
* Severe esophagitis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Weight loss | 48 weeks
  Weight in Kg and Body Mass Index (BMI) in kilograms by meters squared

SECONDARY OUTCOMES:
Blood count | 48 weeks
  Measured in cmm
Hb1AC | 48 weeks
  Measured in percentage
Cholesterol | 48 weeks
  Measured in mg/dL
Fasting blood glucose | 48 weeks
  Measured in mg/dL
Procedural complications | At the time of procedure and at 6 months and 1 year follow-up period
  Complications related to the procedure, either at the time of the procedure (bleeding, perforation and suture rupture) or in the postoperative period, performing an endoscopy at 6 months and 1 year to evaluate the suture line.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Guatavo de Quadros, MD, Principal Investigator — Kaiser Clinica and Day Hospital
Locations (3):
- Brazil (3):
  - Mario Covas Hospital, Santo André, São Paulo
  - Kaiser Day hospital, São José do Rio Preto, São Paulo
  - 9 de Julho Hospital, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes